CLINICAL TRIAL: NCT04123964
Title: Use of Probabilist Broad-spectrum β-lactam for One-stage Replacement of Infected Hip / Knee Arthroplasties: Retrospective Analysis in a Center of Reference
Brief Title: β-lactam Use in Single-stage Exchange of ProstheTic Infections (Knee / Hip) in a Center of Reference (β-SEPTIC)
Acronym: β-SEPTIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7368
Record Dates: First submitted 2019-09-27; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-09

CONDITIONS: Infected of Hip or Kneeprosthesis
Keywords: Peri-prosthetic infection; Joint infection; One-stage replacement; Broad-spectrum β -lactam

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to the official recommendations, infected prosthesis can be surgically treated by one or two-stage replacement. In Strasbourg, the investigators only perform one-stage surgery, which means that the new materiel is put directly into an infected site. To prevent re-infection, probabilist antibiotherapy has to be started the earlier as possible and to have the larger specter as possible. Official recommendations don't specify the best choice of antibiotherapy and let prescriptors make choice, according to the local epidemiology and patient's history.

In Strasbourg, the investigators systematically start an antibiotic against cocci gram positive: daptomycin. Sometimes, the investigators add tazocillin, a broad-spectrum β-lactam against bacillus gram negative. To determine if the investigators use the second one, they focalized on the presence of fistula or not. Indeed, enterobacteriae from gastro-intestinal tractus are also found on the skin and can move to the peri-prosthetic site if a fistula is created. The major disadvantage of this board-spectrum antibiotic is the selection and creation of resistant bacteriae, which can be responsible of failure, re-infection, or just spreading on the environnement.

The primary purpose is to evaluate retrospectively the prescription of tazocillin, judging it's necessity thanks to antibiograms performed on samples taken during surgery. The aim is to evaluate if the criteria " fistula or not " is a good one to guide the prescription of board-spectrum β-lactam.

Secondary purposes are to find the etiology of failures ( bacteriological failure or re-infection with a new pathogen), evaluate the apparition of multi-drug resistant bacteriae and infections they are responsible for, looking for others criterias which could help the investigators to choose the probablist antibiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Adults ( > 18 years-old) hospitalized from 1st January 2018 to 31th December 2018 in the septic orthopedic surgery unity of the university hospital of Strasbourg for a prosthetic-joint infection (knee or hip) treated by replacement.
* Patients who mentioned they agree for scientific use of their medical data.

Exclusion Criteria:

* Patients hospitalized only for the second surgery of a two-stage replacement.
* Patients who refused or didn't agree with scientific use of their medical data.
* Adults with legal protective measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ( > 18 years-old) hospitalized from 1st January 2018 to 31th December 2018 in the septic orthopedic surgery unity of the university hospital of Strasbourg for a prosthetic-joint infection (knee or hip) treated by replacement
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of the use of β-lactams in infected of hip or knee prosthesis | Files analysed retrospectily from January 1st, 2018 to December 31st, 2018 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Orthopédique Septique, Strasbourg, France